CLINICAL TRIAL: NCT04128397
Title: An Exploratory Study of Continuous Theta Burst Stimulation (cTBS) Based on Functional Magnetic Resonance Imaging (fMRI) in the Treatment of Tic Disorder
Brief Title: An Exploratory Study of Continuous Theta Burst Stimulation (cTBS) Based on fMRI in the Treatment of Tic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20181207
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-06

CONDITIONS: Tic Disorders; Tourette Syndrome
Keywords: continuous theta burst stimulation (cTBS); fMRI
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: first group is traditional stimulation site group ,second group is precise position stimulation group .
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional stimulation site continuous theta burst stimulation (cTBS) (Experimental): arm: experimental: performing cTBS to tic patients for continuous 5 days ,3 times for a day (0 minute ,15 minute ,60 minute). The stimulation site include left supplementary motor area, right supplementary motor area, left primary motor area, right primary motor area , left superior parietal lobule, right superior parietal lobule. Determination of stimulation target is a common method of determination in previous studies. For example the vertex (Cz) was measured for each patient and the SMA defined at 15% of the distance between inion and nasion anterior to Cz on the sagittal midline.
  Interventions: Device: traditional stimulation site continuous theta burst stimulation (cTBS)
- precise stimulation site cTBS (Experimental): arm: experimental: performing cTBS to tic patients for 5 days ,3 times for a day (0 minute ,15 minute ,60 minute). The stimulation site include left supplementary motor area, right supplementary motor area, left primary motor area, right primary motor area , left superior parietal lobule, right superior parietal lobule. The stimulation target is determined by the resting-state functional connectivity, which is robust functional connectivity with the GPi or Thalamus.
  Interventions: Device: precise stimulation site cTBS

INTERVENTIONS:
Device: traditional stimulation site continuous theta burst stimulation (cTBS) — before cTBS treatment, MRI was used to confirm the stimulation site
  Arms: traditional stimulation site continuous theta burst stimulation (cTBS)
Device: precise stimulation site cTBS — before cTBS treatment, rs-fMRI was used to confirm the stimulation site
  Arms: precise stimulation site cTBS

SUMMARY:
continuous theta burst stimulation (cTBS) is a safe and effective device for Gilles de la Tourette's syndrome treatment. GPi is an agreed curative target of deep brain stimulation. GPi-based functional connectivity peak voxel in the SMA can be the cTBS target.

DETAILED DESCRIPTION:
Tic disorder is a common neuropsychiatric disorder in children and adolescents. Medication is not effective and has side effect. Exploring new treatment methods is one of the research pathway of this disease.Continuous theta burst stimulation (cTBS) is relatively safe and effective, and its efficacy in psychiatric diseases has been gradually recognized. However, the results of current researches of tic disorder treatment are varied, and the evaluation method is relatively single. This project intends to adopt fmri-guided stimulation target and navigated cTBS to intervene patients with tics and explore individualized cTBS treatment parameters of tics, including stimulation frequency, intensity, type, time and stimulation target. Previous studies for deep brain stimulation reported that the medial globus pallidus (GPi) showed an obvious curative effect. And a deep brain area can be modulated indirectly by a superficial target via functional connectivity. Therefore, the present study attempts to stimulate the superficial target in supplementary motor area (SMA), lateral motor area (M1) which functionally connected with GPi or thalamus since the thalamus also a commonly reported abnormal brain area of Tic. Combined with clinical symptoms and neuroimaging, the therapeutic effect of cTBS in children with tic disorder was comprehensively evaluated in order to provide a new therapeutic method and a better therapeutic effect for the disease.

ELIGIBILITY:
Inclusion Criteria:

1. meet the diagnostic criteria of chronic tic disorder or tourette syndrome;
2. Yale Global Tic Severity Scale (YGTSS) score is greater than 20;
3. the symptoms lasted more than 1 year, and the drug regimen was not adjusted within one month;
4. right-handedness;
5. age 6-20 years;
6. able to receive continuous theta burst stimulation (cTBS) therapy, participants and their guardians agree to receive treatment and observation.

Exclusion Criteria:

1. age is under 6-year old;
2. can not tolerate MRI or cTBS treatment;
3. adjust medication during treatment.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale score | 5 days
  to evaluate clinical change

SECONDARY OUTCOMES:
fMRI | 1 day, 5 days
  local neural activity; functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Feng, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - center for cognition and brain disorders,HZNU, Hangzhou, Zhejiang
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grados M, Huselid R, Duque-Serrano L. Transcranial Magnetic Stimulation in Tourette Syndrome: A Historical Perspective, Its Current Use and the Influence of Comorbidities in Treatment Response. Brain Sci. 2018 Jul 6;8(7):129. doi: 10.3390/brainsci8070129. PMID 29986411
- [Background] Landeros-Weisenberger A, Mantovani A, Motlagh MG, de Alvarenga PG, Katsovich L, Leckman JF, Lisanby SH. Randomized Sham Controlled Double-blind Trial of Repetitive Transcranial Magnetic Stimulation for Adults With Severe Tourette Syndrome. Brain Stimul. 2015 May-Jun;8(3):574-81. doi: 10.1016/j.brs.2014.11.015. Epub 2014 Dec 3. PMID 25912296
- [Background] Johnson KA, Fletcher PT, Servello D, Bona A, Porta M, Ostrem JL, Bardinet E, Welter ML, Lozano AM, Baldermann JC, Kuhn J, Huys D, Foltynie T, Hariz M, Joyce EM, Zrinzo L, Kefalopoulou Z, Zhang JG, Meng FG, Zhang C, Ling Z, Xu X, Yu X, Smeets AY, Ackermans L, Visser-Vandewalle V, Mogilner AY, Pourfar MH, Almeida L, Gunduz A, Hu W, Foote KD, Okun MS, Butson CR. Image-based analysis and long-term clinical outcomes of deep brain stimulation for Tourette syndrome: a multisite study. J Neurol Neurosurg Psychiatry. 2019 Oct;90(10):1078-1090. doi: 10.1136/jnnp-2019-320379. Epub 2019 May 25. PMID 31129620